CLINICAL TRIAL: NCT00885534
Title: Genetic Variates of Response to Cisplatin, Vinblastine, and Temozolomide (CVT) in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-017
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Results first posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Melanoma; Skin Cancer
Keywords: skin cancer; CISPLATIN; TEMOZOLOMIDE; VINBLASTINE; 09-017
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Cisplatin; Vinblastine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemotherapy (Experimental): This is a single institution phase II trial in stage III or IV melanoma patients with measurable disease but no prior cytotoxic chemotherapy and not thought to be curable by surgery.Before starting the chemotherapy, you may need to have a fresh biopsy of your tumor. If you have already had a tumor biopsy that we can use, you may not need another biopsy. Your study doctor will review with you the biopsies you have had. We will try to obtain biopsy material that already exists but if we cannot, you will need another biopsy.
  Interventions: Drug: Cisplatin, Vinblastine, Temozolomide

INTERVENTIONS:
Drug: Cisplatin, Vinblastine, Temozolomide — Patients will receive CVT chemotherapy which consists of the following:
  Cisplatin 25 mg/m2 given intravenously on days 2-5 Vinblastine 1.5 mg/m2 given as an intravenous push on days 2-5 Temozolomide 150 mg/m2 given orally on days 1-5. In patients who cannot receive temozolomide, dacarbazine can be used instead. Dacarbazine will be given at 800 mg/m2 IV on day 1.

SUMMARY:
The investigators want to learn to predict which tumors will respond to CVT chemotherapy. CVT is a combination of three drugs - cisplatin, vinblastine, and temozolomide. We and other investigators have used CVT in melanoma patients and found that tumors got significantly smaller in 30-40% of cases. In this study, the investigators want to get a precise idea of how many patients will respond to CVT. Also they want to test which genes in the tumor are turned on and which are turned off. We hope this will teach us to know in the future which tumors will respond to CVT.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologic proof of melanoma reviewed and confirmed at MSKCC
* Patients must have stage IV melanoma or recurrent stage IIIb or IIIc melanoma. Patients who are potentially respectable will be eligible.
* Measurable disease (RECIST criteria). Patients must have a tumor amenable to biopsy for oligonucleotide microarray analysis and for immunohistochemistry. A pre-treatment biopsy is required; a fine needle aspirate is not adequate.
* No prior cytotoxic chemotherapy for melanoma. Prior immunotherapy or anti-angiogenic therapy is allowed.
* No other concurrent chemotherapy, immunotherapy, or radiotherapy
* ECOG performance status ≤ 1
* Adequate organ function defined as follows: ANC >1500/mm3, Platelets >130,000/mm3, calculated creatinine clearance ≥60 ml/minute (Cockcroft & Gault).
* Adequate cardiac function to tolerate the hydration needed for cisplatin administration.

Exclusion Criteria:

* History of CNS metastases unless brain metastases have been resected or successfully treated with stereotactic radiosurgery and the patient has been free from CNS recurrence for 3 months.
* Uveal melanoma primary
* Patients who have had prior anti-CTLA4 monoclonal antibody treatment must have been off treatment for at least 4 months and have signs of progression of disease.
* Frequent vomiting or medical conditions that could interfere with oral medication intake
* Serious infection requiring antibiotics, or nonmalignant medical illnesses that are uncontrolled or whose control might be jeopardized by the complications of this therapy.
* History of HIV infection even if on HAART
* Immunosuppressive drugs
* High dose vitamins and herbs
* Other on-going investigational therapy, concurrent chemotherapy, immunotherapy or radiotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chapman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cisplatin, Vinblastine, Temozolomide
Started | 7
Completed | 6
Not Completed | 1
Not completed — Patient deemed ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin, Vinblastine, Temozolomide
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Response to CVT Chemotherapy.
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Cisplatin, Vinblastine, Temozolomide
Number analyzed (Participants) | 6
participants
  Partial Response | 1
  Stable Disease | 5

ADVERSE EVENTS:
Arm/Group | Cisplatin, Vinblastine, Temozolomide
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin, Vinblastine, Temozolomide (N=6)
Constipation (Gastrointestinal disorders) | 1 (2)
Dehydration (General disorders) | 2 (2)
Hypotension (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin, Vinblastine, Temozolomide (N=6)
Creatinine increased (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Urogenital disorder (Renal and urinary disorders) | 1 (1)
ALT, SGPT (Blood and lymphatic system disorders) | 1 (1)
Fever (in the absence of neutropenia) (General disorders) | 1 (1)
Glucose, high (hyperglycemia) (General disorders) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 2 (2)
Potassium, high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Bilirubin (hyperbilirubinemia) (Blood and lymphatic system disorders) | 1 (1)
INR increased (Blood and lymphatic system disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes